CLINICAL TRIAL: NCT00821210
Title: Obstructive Sleep Apnea and Acute Myocardial Infarction and the Role of CPAP Treatment: a Double -Blind, Randomized Control Trial
Brief Title: Obstructive Sleep Apnea and Acute Myocardial Infarction and the Role of Continuous Positive Airway Pressure (CPAP)Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Peilin Lee, National Taiwan University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200712052R
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Sleep Apnea, Obstructive; Acute Myocardial Infarction
Keywords: Obstructive sleep apnea; myocardial infarction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Sham Comparator)
  Interventions: Device: Sham CPAP
- 1 (Active Comparator)
  Interventions: Device: CPAP of optimal pressure

INTERVENTIONS:
Device: Sham CPAP — CPAP with pressure of 3cm H2O
  Arms: 2
Device: CPAP of optimal pressure — CPAP of optimal pressure
  Arms: 1

SUMMARY:
Specific Aim

1. To determine the prevalence of OSA in patients of first-time AMI in acute phase By screening patients of first-time, single-vessel disease, Killip I AMI, and successful revascularization
2. To determine the impact of CPAP treatment on the prognosis of AMI Using sham CPAP as the optimal placebo, we conduct this randomized, double-blind, placebo controlled trial to assess the 12-week CPAP effect in moderate-severe OSA patients.
3. To determine how the OSA affects patients with MI in acute and chronic phase and vice versa, which is dissected from mechanical basis and molecular basis By comparing the clinical parameters of AMI patients without OSA (AHI<5/hr), mild OSA (5 < AHI <15), moderate OSA (15<AHI<30) and severe OSA5 (AHI>30/hr), and before and after CPAP treatment, we can determine the interaction between OSA and AMI.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a major public health problem affecting at least 2-4% of middle-aged population. OSA resulted in hypoxia and sleep fragmentation, which resulted in neurocognitive dysfunction and cardiovascular sequelaes. The cardiovascular sequelaes in OSA included hypertension, coronary artery disease and heart failure. Our data showed among 599 moderate-sever OSA (AHI<15/hr)， 44.5% patients had cardiovascular disease, which included 41.4% having hypertension，7% having CAD and 2.4% having congestive heart failure。 Though OSA is well known to be highly correlated with fatal and non-fatal cardiac event, only limited studies investigated how OSA affected acute myocardial infarction (AMI). Most studies concluded that AMI would worsen OSA and vice versa. However, how AMI exactly interacts with OSA and what the prevalence of OSA in the first-time AMI is have never been answered. Within four weeks from Nov. 15th 2007, we screened ten patients of first-time AMI with single-vessel disease and Killip I. Five in 10 received PSG and three in five have moderate OSA.

So far, CPAP is the standard treatment for patients with moderate to severe OSA. CPAP could improve airway patency, daytime sleepiness, functional status, blood pressure, metabolic abnormalities and quality of life. In our study, we enrolled 24 non-sleepy OSA and 30 sleepy OSA to study the four-week CPAP effect. The results showed the apnea-hypopnea index, hypoxia, arousal, sleepiness and fatigue could be corrected with CPAP treatment in both groups. However, CPAP could only lower risk factors for cardiovascular disease, like blood pressure, epinephrine, norepinephrine and CRP, in sleepy OSA. Our finding supported that CPAP effect was not similar in the subgroups of severe OSA, so CPAP effect should be studied in every subgroup of OSA patients before it's applied. Till now, there's no literatures reported if CPAP treatment would decrease the morbidity and mortality of AMI.

Sham CPAP mimicked all the characteristics of a true CPAP except for the null pressure, which was recently used as the placebo to study CPAP effect. Therefore, using this optimized placebo, we propose this double-blind, control randomized trial (1) To determine the prevalence of OSA in patients of first-time AMI in acute phase; (2) To determine the impact of CPAP treatment on the prognosis of AMI; (3) Determine how the OSA affects patients with MI in acute and chronic phase and vice versa, which is dissected from mechanical basis and molecular basis.

ELIGIBILITY:
Inclusion Criteria:

1. First-time AMI
2. s/p revascularization (successful primary PTCA for ischemia-related artery)
3. Killip I

Exclusion Criteria:

1. Refuse to participate
2. Require mechanical ventilation
3. Having active neurologic event, severe obstructive airway disease and active infection, active malignancy
4. Need sedative drug or narcotics during the study period within 3 days of PSG
5. Participates other study at the same time

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary goal: Intervention: Improvement of LVEF by 7%, decrease the left ventricular end-systolic dimension by 3 mm, 3D echo. | 12 weeks

SECONDARY OUTCOMES:
incidence of stroke and fetal, non-fetal cardiac event | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jen Yu, M.D., Principal Investigator — National Taiwan University Hospital; Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan